CLINICAL TRIAL: NCT01783132
Title: Optimization of Inhaled Corticosteroid Treatment in Adult Patients With Asthma Guided by Exhaled NO Measurement at Home
Acronym: OCTAGEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changing conditions for the device in one of the participation companies
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1852011
Record Dates: First submitted 2013-01-11; First posted 2013-02-04 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: SOC
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Other): Asthma treated patient with Budesonide for 1 year, 4 different dosage according to measurement of exhaled NO done with NIOX MINO.
  Interventions: Device: NIOX MINO
- Standard of care (No Intervention): Asthma treated patient with standard of care during 1 year. Exhaled NO measurement will be done 4 times/year, and compared afterwards with the Budesonide group.

INTERVENTIONS:
Device: NIOX MINO — Active group (Budesonide) will be measuring exhaled NO at least 3 times/week at home to control their Asthma treatment via a algorithm schedule. The control group (Standard of care) will be measuring exhaled NO 4 times/year at study site.
  Arms: Budesonide

SUMMARY:
To compare the clinical outcome (effectiveness) of single inhaled corticosteroid (ICS) controller treatment guided by exhaled NO measurement made at home with usual care asthma management with regard to asthma control (primary outcome), asthma-related quality of life, lung function, airway inflammation, medication use, and asthma events.

To understand changes in patient behaviour triggered by daily FENO measurement at home, for example treatment adherence and voluntary allergen exposure.

DETAILED DESCRIPTION:
The design is a pragmatic randomized controlled, open-label, parallel group study Screening visit 1 and visit 2 is separated with a 2-4 week run-in period. At screening visit, Informed Consent is signed and atopic asthma confirmed, spirometry is performed and questionnaires responded to. At visit 2 venous blood samples are taken and serum stored at -20 °C for later transport to Uppsala Biobank, Exhaled NO is measured at both visit using NIOX MINO (blinded in control group).

* The active group if on combination inhaler, will switch to Giona Easyhaler (same budesonide equivalent as before study entry) and Oxis (same formoterol equivalent as before study entry). These patients will receive a NIOX MINO and will be taught about the adjustment of ICS treatment according to daily exhaled NO measurement at home and a personalized treatment algorithm.
* The control group will stay on previous controller treatment (only changed if indicated by symptoms at visit) according to usual care.
* Both groups will switch short-acting beta-2-agonist to Buventol Easyhaler.
* Both groups will report symptoms (ACQ) monthly and in connection to asthma events via an ePRO system (ViedocMe, PCG). Active group will report NO values on a weekly basis via the same system.

There will be a follow-up clinic visit 3 at 6 months with exhaled NO measurement (blinded in control group) and limited set of questionnaires. A second follow-up visit 4 at 12 months with exhaled NO, spirometry, full set of questionnaires and blood sample will be made.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, ≤64 years
* Physician-diagnosis of asthma
* Regular inhaled budesonide (Giona Easyhaler, Pulmicort Turbuhaler, Novopulmon Novolizer or Symbicort Turbuhaler) treatment since at least 6 months
* Verified allergy to at least one airborne perennial allergen after objective testing (ImmunoCAP Rapid Asthma/Rhinitis Adult)
* ACQ >1.0
* Can read and understand the Swedish language
* Written informed consent signed

Exclusion Criteria:

* Regular tobacco use within past 6 months
* ≥10 pack-years smoking history
* Keeping a furred pet at home
* Treatment with Singulair
* >4 prednisolone courses last 12 months
* Ongoing pregnancy or lactation
* Participation in another clinical trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-28 (Actual)

PRIMARY OUTCOMES:
Asthma symptoms in correlation to grade of inflammation in airways | Up to 1 year
  To determine if ICS treatment guided by daily FENO measurement with a device "NIOX MINO" at home will improve asthma symptom control compared to usual care asthma management

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Alving, Dr, Study Director — Aerocrine AB
Locations (1):
- Lungkliniken, Universitetssjukhuset i Uppsala, Uppsala, Sweden